CLINICAL TRIAL: NCT05191290
Title: Comparison of Biocompatibility of Plasmapheresis Procedures With Citrate and Heparin Anticoagulation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Jakob Gubensek, Principal investigator, University Medical Centre Ljubljana
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0120-310/2017/3
Record Dates: First submitted 2021-12-12; First posted 2022-01-13 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Apheresis; Anticoagulation
MeSH Terms: interventions — Heparin; Sodium Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- heparin anticoagulation (Active Comparator): standard heparin anticoagulation during plasmapheresis
  Interventions: Drug: unfractionated heparin
- citrate anticoagulation (Experimental): sodium citrate anticoagulation during plasmapheresis
  Interventions: Drug: Sodium Citrate

INTERVENTIONS:
Drug: unfractionated heparin — standard heparin at 2500 IU i.v. bolus and then 2000 IU/h continuously i.v. for anticoagulation during plasmapheresis
  Arms: heparin anticoagulation
Drug: Sodium Citrate — 8% sodium citrate at approx. 27 mmol/h i.v. for anticoagulation during plasmapheresis
  Arms: citrate anticoagulation

SUMMARY:
Membrane plasmapheresis is one of the methods for treating immune diseases. Plasmapheresis removes autoantibodies and immune complexes, paraproteins, lipoproteins and reduces the concentration of cytokines. In membrane plasmapheresis, plasma is separated from blood cells by a highly permeable membrane. The filtered plasma is then discarded and replaced with replacement fluid. During the procedure, there is an activation of the coagulation system, because of the extracorporeal blood circulation. The anticoagulation during the procedure is therefore necessary.

DETAILED DESCRIPTION:
Standard heparin or citrate is routinely used as a method of anticoagulation in plasmapheresis. Citrate provides effective anticoagulation that is completely limited to extracorporeal circulation. Patients who are at increased risk for bleeding, anticoagulation with citrate is a more appropriate method than standard heparin, while in other patients both methods are equivalent.

Citrate anticoagulation is performed by infusing citrate into the arterial line of the extracorporeal system. Citrate binds to plasma calcium and thus inhibits coagulation in the system. Calcium is added to the venous line of the system (when blood returns to the patient) to maintain a normal plasma ionized calcium concentration. Lowering the ionized calcium in the blood in the extracorporeal circulation inhibits the coagulation and activation of other systems (platelets, leukocytes, complement), which affects the biocompatibility of the artificial material and the whole procedure. Biocompatibility is extremely important, since the contact of blood with artificial material activates both the humoral and cellular systems. As part of the humoral immune system, complement is activated by the production of C3, C4 and C5, factor XIIa, there is also an increase in the production of bradykinin, kallikrein, quinine and plasmin, and some proteins are denatured (gamma globulins, fibrinogen, albumins). When the cellular immune system is activated, lymphocytosis can occur and the is also change in function of phagocytes.

All previous studies show that regional anticoagulation with citrate improves biocompatibility in hemodialysis procedures (compared to heparin anticoagulation), but no direct comparison in plasmapheresis has been observed in the literature so far.

Therefore, the investigators want to conduct a prospective randomized study comparing several parameters of heparin and citrate anticoagulation biocompatibility during plasmapheresis. The aim of the study is to demonstrate better biocompatibility in citrate anticoagulation compared to heparin.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years
* an indication for plasma exchange (plasmapheresis) with albumin solution as a replacement solution

Exclusion Criteria:

* contraindication for systemic heparinisation
* acute bleeding
* known active malignancy
* severe infection
* anticoagulant therapy at therapeutic dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
change in serum thrombin-antithrombin complex from baseline to 30 minutes | 30 minutes after start of plasmapheresis
  thrombin-antithrombin complex
change in serum thrombin-antithrombin complex from baseline to the end of plasmapheresis | at the end of plasmapheresis procedure
  thrombin-antithrombin complex
change in serum platelet factor 4 from baseline to 30 minutes | 30 minutes after start of plasmapheresis
  platelet factor 4
change in serum platelet factor 4 from baseline to the end of plasmapheresis | at the end of plasmapheresis procedure
  platelet factor 4
change in serum C5a from baseline to 30 minutes | 30 minutes after start of plasmapheresis
  complement component C5a
change in serum C5a from baseline to the end of plasmapheresis | at the end of plasmapheresis procedure
  complement component C5a
change in serum myeloperoxidase from baseline to 30 minutes | 30 minutes after start of plasmapheresis
  myeloperoxidase
change in serum myeloperoxidase from baseline to the end of plasmapheresis | at the end of plasmapheresis procedure
  myeloperoxidase

SECONDARY OUTCOMES:
complications during plasmapheresis (hypocalcemia, metabolic alkalosis, clotting) | during plasmapheresis
  complications during plasmapheresis (hypocalcemia, metabolic alkalosis, clotting)
comparison of measured platelet factor 4 in patients' serum and filtered plasma | 30 minutes after start of plasmapheresis
  A Bland-Altman agreement analysis
comparison of measured thrombin-antithrombin complex in patients' serum and filtered plasma | 30 minutes after start of plasmapheresis
  A Bland-Altman agreement analysis
comparison of measured C5a in patients' serum and filtered plasma | 30 minutes after start of plasmapheresis
  A Bland-Altman agreement analysis
comparison of measured myeloperoxidase in patients' serum and filtered plasma | 30 minutes after start of plasmapheresis
  A Bland-Altman agreement analysis

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No